CLINICAL TRIAL: NCT02602158
Title: The13C Trioctanoate Breath Test as a Measurement Method for the Gastric Emptying of Fat; a Randomised, Single Blinded, Cross Over Study
Brief Title: 13C Trioctanoate Breath Test as a Measurement of Gastric Fat Volume Emptying
Acronym: 13CTriOBT
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: KEK-Nr. 2015-0450
Record Dates: First submitted 2015-10-28; First posted 2015-11-11 (Estimated); Last update posted 2016-07-22 (Estimated); Status verified 2016-07

CONDITIONS: Healthy
Keywords: breath test; lipid emulsions; MRI; gastric emptying
MeSH Terms: interventions — octanoic acid; tricaprylin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Octanoic acid (1-13C, 99%) (Active Comparator): 100 µL 13C Octanoic acid (Cambridge isotope laboratories)
  Interventions: Dietary Supplement: Octanoic acid (1-13C, 99%)
- TRIOCTANOIN (1,1,1-13C3, 99%) (Active Comparator): 100 µL 13C Trioctanoin (Cambridge isotope laboratories)
  Interventions: Dietary Supplement: TRIOCTANOIN (1,1,1-13C3, 99%)

INTERVENTIONS:
Dietary Supplement: Octanoic acid (1-13C, 99%) — 13C-marker will be mixed with emulsions. 2 isovolumetric (200 ml) and isocaloric (200 kcal) lipid emulsions with different acid and shear stability Lipid emulsion 1: acid stable, particle size 0.6 µm
  Optional study pending interim analysis:
  Lipid emulsion 4: acid unstable, redispersible by mechanical processes during antral contractions and passage through the pylorus, particle size 0.6 µm
  Arms: Octanoic acid (1-13C, 99%)
Dietary Supplement: TRIOCTANOIN (1,1,1-13C3, 99%) — 13C-marker will be mixed with emulsions 2 isovolumetric (200 ml) and isocaloric (200 kcal) lipid emulsions with different acid and shear stability
  Lipid emulsion 1: acid stable, particle size 0.6 µm
  Optional study pending interim analysis:
  Lipid emulsion 4: acid unstable, redispersible by mechanical processes during antral contractions and passage through the pylorus, particle size 0.6 µm
  Arms: TRIOCTANOIN (1,1,1-13C3, 99%)

SUMMARY:
13C breath tests represent an attractive alternative in the measurement of gastric emptying (GE). Therefore these tests have been used in a variety of clinical settings such as in the assessment of gastroparesis, delayed GE in diabetic patients or in the assessment of GE with fat containing enteral formulas in critically ill patients.

The investigators have previously demonstrated that the 13C sodium octanoate breath test (OBT) is an inappropriate measurement method for the GE of fat. The OBT appears to be affected by 1) post gastric processing of the OCC marker and 2) its interaction with the physical form and concentration of the fat present in the stomach and duodenum.

The13C trioctanoate breath test (TriOBT) represents an attractive alternative to the OBT. Compared to OCC which is a medium chain fatty acid the 13C trioctanoate (TriOCC) is a triglyceride. TriOCC has similar physio chemical properties as the nutritional lipid e.g. rapeseed oil.

This study aims to assess the efficacy of the TriOBT as a GE measurement method of fat in an acid stable lipid emulsion (LE1). The breath test results from the TriOBT will be compared with the OBT and further validated against gastric fat volume emptying data observed from MRI. The interim analysis will determine whether the study will proceed to stage 2 which will assess the efficacy of the TriOBT in an acid unstable lipid emulsion (LE4).

DETAILED DESCRIPTION:
13C breath tests for the measurement of gastric emptying (GE) were first developed in the early 1990s. These tests have clear advantages over many other GE imaging techniques as they are relatively inexpensive, simple to use, can be carried out in children and pregnant women or those who have contraindications to MRI. Therefore these tests have been used in a variety of clinical settings such as in the assessment of gastroparesis or delayed GE in diabetic patients or the assessment of GE with fat containing enteral formulas in critically ill patients. Breath tests rely upon the ingestion of a 13C stable isotope markers such as the medium chain fatty acid 13C octanoic acid (OCC) and the tryglyceride13C trioctanoate (TriOCC).

However, 13C breath tests are an indirect measure of GE. Thus, GE data acquired from breath tests are a result of numerous complex interactions which include: 1) the chemical properties of markers and their interactions with test meals during gastric processing 2) absorption from the duodenum, 3) metabolism by the liver (oxidation of fatty acids) and 4) final excretion as 13CO2 by the lungs. All of these complex interactions can become compounded when the gastric processing of lipid emulsions (LEs) are investigated and thus careful consideration and selection of breath test markers is required.

The investigators have developed isocaloric and isovolume LEs with different GE properties as shown previously with MRI. The acid stable (LE1) and acid unstable lipid emulsion (LE4) responds differently to the conditions within the stomach. LE1 empties relatively uniformly from the stomach. However, the LE4 separates into water and high fat phases after 15-30 min of being in the stomach. In the late phase of GE the emulsion is re-emulsified and thus there are three distinct GE phases in LE4. Once separation of LE4 occurs the aqueous and low fat phase empties fairly rapidly from the stomach whereas the second fat phase empties more slowly. The differing GE pattern of acid unstable LEs has a profound effect on GE breath test data dependent upon the selection of the breath test marker used.The investigators have previously demonstrated that the OCC breath test (OBT) is an inappropriate measure of the gastric emptying of fat as the OBT is influenced by 1) Post gastric processing of the OCC marker and 2) its interaction with the physical form and concentration of the fat present in the stomach and duodenum. These effects were highlighted by only a marginal concordance agreement with the OBT half emptying (T50) of 13CO2 recovery and fat volume T50 (MRI T50) with LE1 and no agreement with LE4 (rc=0.7 and rc=0.4 respectively)..

The main aim of this study is to investigate whether TriOCC is a more appropriate breath test marker to use in the measurement of the GE of fat. As the TriOCC is a triglyceride it has similar physiochemical properties to nutritional lipids. Therefore, it is more likely to behave similarly in the gastric and duodenal environment to ingested lipids in emulsions such as rapeseed oil. In study 1 the investigators will compare the breath test markers TriOCC and OCC in LE1. In a sub set of participants a validated MRI quantitative fat fraction method will be used to determine reference values for the half gastric emptying time of fat (MRI T50). This will be correlated to half emptying (T50) of 13CO2 recovery generated from percentage dose recovery per hour (PDR/h) curves. The interim analysis will assess whether the TriOCC is more related to gastric fat volume emptying than the OCC marker in LE1. Should TriOCC be representative of gastric fat volume emptying study 2 will then proceed. Study 2 will then assess the gastric emptying of fat as above but with LE4.

A secondary aim is to develop an algorithm to quantify the heterogeneity of fat distribution within gastric content for MRI data. The gastric processing of lipid emulsions as visualized by MRI has been shown to result in a large inter individual variation of fat distribution. By quantifying this heterogeneity we aim to determine the degree of flocculation and creaming of the emulsions across the length of the stomach.

ELIGIBILITY:
Inclusion Criteria:

* BMI 18-25 kg/m²
* Written informed consent
* 18 Years to 50 Years

Exclusion Criteria:

* History of GI, cardiorespiratory (including arterial
* hypertension), hematologic, renal, atopic, alimentary or psychiatric disorder, panic attacks, diabetes
* Prior abdominal surgery other than uncomplicated appendectomy or hernia repair
* Requiring medication that might alter gut function, including calcium channel blockers, prokinetics, macrolide antibiotics
* Presence of metallic implants, devices or metallic foreign bodies
* Pregnancy and lactation (female participants of child bearing age will receive a pregnancy test prior to study)
* Claustrophobia
* Regular smoking
* A history of drug or alcohol abuse
* A history of food allergies or intolerances
* Uncertainty about the willingness or ability of the participant to comply with the protocol requirements

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2015-10; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Half emptying time (T50) [min] as determined from 13CO2 recovery curves in breath using the exponential beta function | upto 300 min

SECONDARY OUTCOMES:
The T50 [min] of MRI fat volume emptying | up to 180 min
Correlation of MRI T50 [min] and breath test T50 [min | up to 180 min (MRI) and every 10 min until 300 min (breath test)
The maximum secretion volume [ml] | up to 180 min
Spatial heterogeneity of gastric content will be assessed using a variogram approach | up to 180 min

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Steingötter, PhD, Principal Investigator — Univeristy of Zürich
Locations (1):
- University Hopsital Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Parker HL, Liu D, Curcic J, Ebert MO, Schwizer W, Fried M, Steingoetter A. Gastric and Postgastric Processing of 13C Markers Renders the 13C Breath Test an Inappropriate Measurement Method for the Gastric Emptying of Lipid Emulsions in Healthy Adults. J Nutr. 2017 Jul;147(7):1258-1266. doi: 10.3945/jn.117.248765. Epub 2017 May 31. PMID 28566523
- [Derived] Liu D, Parker HL, Curcic J, Kozerke S, Steingoetter A. Emulsion Stability Modulates Gastric Secretion and Its Mixing with Emulsified Fat in Healthy Adults in a Randomized Magnetic Resonance Imaging Study. J Nutr. 2016 Oct;146(10):2158-2164. doi: 10.3945/jn.116.234955. Epub 2016 Sep 7. PMID 27605407